CLINICAL TRIAL: NCT04958603
Title: The Clinical Effect of Different Lateral Retinaculum Relaxation Methods in the Treatment of Lateral Patellar Compression Syndrome
Brief Title: The Clinical Effect of Different Lateral Retinaculum Relaxation Methods in the Treatment of LPCS
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020506
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Lateral Patellar Compression Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional surgery group: Traditionally loosen the lateral support belt proximally
- New surgery group: Laterally loosen the outer support belt, that is, "L"-shaped loosen
  Interventions: Procedure: "L" type release surgery

INTERVENTIONS:
Procedure: "L" type release surgery — Lateral release of the lateral support belt
  Groups: New surgery group

SUMMARY:
To observe the comparison of the clinical effects of two different ways of loosening the lateral support band under arthroscopy to treat lateral patella excessive compression syndrome.

DETAILED DESCRIPTION:
To analyze the surgical conditions of 64 patients with lateral patella excessive compression syndrome who were surgically treated by Deputy Chief Physician Yang Yuping of the Department of Sports Medicine, Peking University Third Hospital from September 2004 to January 2019. Among them, 24 early cases used the traditional proximal release of the lateral retinaculum (traditional surgical group), and recently 40 cases, after learning from the surgical experience of the early cases, switched to the lateral release of the lateral retinaculum, that is, "L" type Release (new surgery group). The visual analog scale (VAS), Lysholm score, and IKDC knee function subjective evaluation scale (IKDC) score were performed before and after the operation. By analyzing the knee movement scores of patients before and after surgery, the efficacy of the above two operations was judged, and the two groups of postoperative scores were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* From September 2004 to January 2019, patients with lateral patella overcrowding syndrome treated by deputy chief physician Yang Yuping of the Department of Sports Medicine, Peking University Third Hospital

Exclusion Criteria:

* From September 2004 to January 2019, patients with lateral patella overcrowding syndrome treated by deputy chief physician Yang Yuping of the Department of Sports Medicine, Peking University Third Hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From September 2004 to January 2019, patients with lateral patella overcrowding syndrome treated by deputy chief physician Yang Yuping of the Department of Sports Medicine, Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | Six months after surgery
  VAS is used to evaluate knee function. The higher the score of VAS, the better the recovery of knee function
(International Knee Documentation Committee) IKDC knee function subjective evaluation form score | Six months after surgery
  IKDC score is used to evaluate knee function. The higher the score of IKDC score, the better the recovery of knee function

CONTACTS AND LOCATIONS:
Overall Officials: yuping yang, Study Chair — Peking University Third Hospital
Locations (1):
- Peking Univerisity Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No